CLINICAL TRIAL: NCT06726317
Title: The Prevalence and Associated Factors of Psychological Distress, and Effectiveness of a 'life Situation Improving Intervention' Among Oral Cancer Patients Attending Tertiary Care Hospitals in the Colombo District
Brief Title: Early Palliative Care for Patients with Oral Cancer in Sri Lanka
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colombo (Other)
Responsible Party: Principal Investigator, Nadisha Ratnasekera, Principal investigator, University of Colombo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC-18 097
Record Dates: First submitted 2024-11-08; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Oral Cancer; Palliative Supportive Care; Psychological Distress; Quality of Life of Patients
Keywords: early palliative care interventions; oral cancer; head and neck cancer; quality-of-life; psychological distress; supportive care; mindfulness therapy
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This was a Quasi Experimental study with a parallel control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group receiving the novel early palliative care package (Experimental): This group received the novel early palliative care intervention package
  Interventions: Behavioral: Early palliative care integration
- Control group (No Intervention): This group received only the existing standard care in the health system and did not receive any special intervention through this study

INTERVENTIONS:
Behavioral: Early palliative care integration — The early palliative care intervention package was developed following the guidelines provided by the UK Medical Research Council for the development of complex interventions. The early palliative care intervention for patients with oral cancer had six components: 1) providing information, 2) addressing acute and functional issues, 3) nutritional care, 4) psychological support, 5) mindfulness therapy, and 6) coordination of the financial allowance. The package was formulated by triangulating literature review findings and several independent studies: a case-control study; in-depth interviews with experts in the field of oncology and palliative care in Sri Lanka; key-informant interviews with patients with oral cancer and their caregivers; and an observation study at the National Cancer Institute Sri Lanka- Apeksha Hospital). The intervention package was finalized through a
  Other Names: Supportive care; Psycho-oncology care
  Arms: Intervention group receiving the novel early palliative care package

SUMMARY:
The goal of this quasi experimental study is to develop and assess the effectiveness of an early palliative care intervention in patients with oral cancer in Sri Lanka. The main question it aims to answer is whether the early palliative care intervention improves the quality of life and psychological distress of patients with cancer in Sri Lanka.

The primary outcome measures were patient's quality of life and level of psychological distress If there is a comparison group: Researchers compared with a control group who received the standard care to see if the novel early palliative care intervention helped to improve the primary outcomes.

Participants in the intervention arm received the early palliative care package which consisted of 6 components including: 1) providing information, 2) addressing acute and functional issues, 3) nutritional care, 4) psychological support, 5) mindfulness therapy, and 6) coordination of the financial allowance. The intervention was delivered by the Principal Investigator and the trained Public Helath Nursing Officers.

DETAILED DESCRIPTION:
The study took place at three tertiary care units providing oral cancer treatment in Sri Lanka: the oral and maxillofacial wards at the National Dental Hospital, Colombo (Teaching); the oral and maxillofacial wards at Colombo South (Teaching) Hospital, Karapitiya; and the onco-surgery wards at the National Cancer Institute Maharagama (Apeksha Hospital).

Participants The study participants were patients with oral cancer whose definitive diagnosis had been communicated to the patient and had psychological distress (score of ≥4 after screening with the Sinhala version of the Distress Thermometer); awaiting surgery as the first treatment modality; and married with children, including at least one family caregiver with the ability to communicate and read well in Sinhalese. Exclusion criteria were, recurrent oral cancer; a formal psychiatric diagnosis; and receiving or having received any early palliative care intervention. They were divided to 55 controls and 55 cases based on the availability of an accessible Public Health Nursing Officer.

Interventions The early palliative care package, comprising six components, was delivered in three sessions by the principal investigator (PI) and Public Health Nursing Officers.

Outcome measures The effectiveness was assessed by the level of psychological distress using the Sinhala version of the Distress Thermometer and Level of quality of life using EORTC QLQ 30 with module H&N 35 at baseline (T0), post-intervention (T1), one month (T2), and three months (T3).

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis communicated to the patient
* Presence of psychological distress (score of ≥4 after screening with the Sinhala version of the Distress Thermometer27)
* awaiting surgery as the first treatment modality
* married with children, including at least one family caregiver with the ability to communicate and read well in Sinhalese.

Exclusion Criteria:

* Recurrent oral cancer
* A formal psychiatric diagnosis
* Receiving or having received any early palliative care intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Patient's quality of life | This outcome measure was collected at four-time points: at enrollment, immediately after delivering the intervention package, 1 month after and three months after the intervention.
  Quality of life was measured using the Sinhala version of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (version C30) -EORTC QLQ 30. This tool was translated and validated to Sri Lanka through a large-scale multi-centre study. This tool measured quality of life in three sub dimensions-Global Health Status, Functional Scale and Symptom Scale. a high score in Global Health Status denoted a high quality of life, a high score for Functional Scale meant healthy level of functioning and a high score in Symptom Scale represented high level of problems
Patient's level of psychological distress | The outcome measures were collected at four-time points: at enrollment, immediately after delivering the intervention package, one month and three months after the intervention.
  The level of psychological distress was measured through the mean scores of the Sinhala version of the Distress Thermometer. The Distress Thermometer is 1 item, an ultra-short, visual analogue screening tool, originally developed in the America for prostate cancer patients in 1998. The Distress Thermometer comes with a Problem List. This has 35 items and it covers 5 life domains (practical, family/social, emotional, spiritual, and physical problems). The Distress Thermometer and Problem List were translated into the Sinhala language (the primary language in Sri Lanka) and cross-culturally adapted to Sri Lanka.
Patient's quality of life related to the Head and Neck condition | This outcome measure was collected at four-time points: at enrollment, immediately after delivering the intervention package, 1 month after and three months after the intervention.
  This was measured using Head & Neck-35 module (H&N-35) by European Organization for Research and Treatment of Cancer. This tool was translated and validated to Sri Lanka through a large-scale multi-centre study. A high score in H&N-35 module also meant high level of problems whcih meant low quality of life.

SECONDARY OUTCOMES:
Patient's satisfaction | This was measured 3 months after the delivery of the intervention package
  Patient's satisfaction with the novel intervention was measured using a validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Irosha Perera, Doctor of Medicine, Study Director — Preventive oral Health Unit, National Dental Hospital, Sri Lanka; Pushpakumara Kandapola Arachchige, Doctor of Medicine, Study Director — National Cancer Institute, Maharagama- Apeksha Hospital, Sri Lanka
Locations (4):
- Sri Lanka (4):
  - Karapitiya Teaching Hospital, Galle, Southern Province
  - National Dental Hospital, Colombo, Western Province
  - Apeksha Hospital, Colombo, Western Province
  - Colombo South (Teaching) Hospital, Colombo, Western Province

IPD SHARING:
Plan to Share IPD: No
IPD will not be required at any level for any purpose. Also, keeping to the ethical conduct- I am obliged to protect the confidentiality of the participants. Therefore, as ICP serve no good purpose I will not share them

REFERENCES:
- [Background] Kadan-Lottick NS, Vanderwerker LC, Block SD, Zhang B, Prigerson HG. Psychiatric disorders and mental health service use in patients with advanced cancer: a report from the coping with cancer study. Cancer. 2005 Dec 15;104(12):2872-81. doi: 10.1002/cncr.21532. PMID 16284994
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Jayasekara H, Rajapaksa LC, Aaronson NK. Health-related quality-of-life in patients with head-and-neck cancer in Sri Lanka: psychometric properties of the 'Sinhala' version of the EORTC QLQ-H&N35. Psychooncology. 2009 Oct;18(10):1116-21. doi: 10.1002/pon.1430. PMID 19142857
- [Background] Jayakar R, Choi J, MacKinnon C, Tan S. The cost of major head and neck cancer surgery. N Z Med J. 2017 May 12;130(1455):111-119. PMID 28494483
- [Background] Jacobsen PB, Jim HS. Psychosocial interventions for anxiety and depression in adult cancer patients: achievements and challenges. CA Cancer J Clin. 2008 Jul-Aug;58(4):214-30. doi: 10.3322/CA.2008.0003. Epub 2008 Jun 16. PMID 18558664
- [Background] Ip WY, Martin CR. Psychometric properties of the 12-item General Health Questionnaire (GHQ-12) in Chinese women during pregnancy and in the postnatal period. Psychol Health Med. 2006 Feb;11(1):60-9. doi: 10.1080/13548500500155750. PMID 17129895
- [Background] Infurna FJ, Gerstorf D, Ram N. The nature and correlates of change in depressive symptoms with cancer diagnosis: reaction and adaptation. Psychol Aging. 2013 Jun;28(2):386-401. doi: 10.1037/a0029775. Epub 2012 Sep 17. PMID 22984800
- [Background] Hutchison SD, Steginga SK, Dunn J. The tiered model of psychosocial intervention in cancer: a community based approach. Psychooncology. 2006 Jun;15(6):541-6. doi: 10.1002/pon.973. PMID 16331595
- [Background] van den Hurk DG, Schellekens MP, Molema J, Speckens AE, van der Drift MA. Mindfulness-Based Stress Reduction for lung cancer patients and their partners: Results of a mixed methods pilot study. Palliat Med. 2015 Jul;29(7):652-60. doi: 10.1177/0269216315572720. Epub 2015 Feb 20. PMID 25701663
- [Background] Humphris GM, Ozakinci G. Psychological responses and support needs of patients following head and neck cancer. Int J Surg. 2006;4(1):37-44. doi: 10.1016/j.ijsu.2005.12.004. Epub 2006 Feb 3. PMID 17462312
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Hopko DR, Bell JL, Armento M, Robertson S, Mullane C, Wolf N, Lejuez CW. Cognitive-behavior therapy for depressed cancer patients in a medical care setting. Behav Ther. 2008 Jun;39(2):126-36. doi: 10.1016/j.beth.2007.05.007. Epub 2007 Oct 31. PMID 18502246
- [Background] Hong JS, Tian J. Sensitivity and specificity of the Distress Thermometer in screening for distress in long-term nasopharyngeal cancer survivors. Curr Oncol. 2013 Dec;20(6):e570-6. doi: 10.3747/co.20.1617. PMID 24311958
- [Background] Holtedahl K, Norum J, Anvik T, Richardsen E. Do cancer patients benefit from short-term contact with a general practitioner following cancer treatment? A randomised, controlled study. Support Care Cancer. 2005 Nov;13(11):949-56. doi: 10.1007/s00520-005-0869-5. Epub 2005 Jul 16. PMID 16025260
- [Background] Holland JC, Bultz BD; National comprehensive Cancer Network (NCCN). The NCCN guideline for distress management: a case for making distress the sixth vital sign. J Natl Compr Canc Netw. 2007 Jan;5(1):3-7. No abstract available. PMID 17323529
- [Background] Holland JC, Andersen B, Breitbart WS, Buchmann LO, Compas B, Deshields TL, Dudley MM, Fleishman S, Fulcher CD, Greenberg DB, Greiner CB, Handzo GF, Hoofring L, Hoover C, Jacobsen PB, Kvale E, Levy MH, Loscalzo MJ, McAllister-Black R, Mechanic KY, Palesh O, Pazar JP, Riba MB, Roper K, Valentine AD, Wagner LI, Zevon MA, McMillian NR, Freedman-Cass DA. Distress management. J Natl Compr Canc Netw. 2013 Feb 1;11(2):190-209. doi: 10.6004/jnccn.2013.0027. PMID 23411386
- [Background] Holland JC. History of psycho-oncology: overcoming attitudinal and conceptual barriers. Psychosom Med. 2002 Mar-Apr;64(2):206-21. doi: 10.1097/00006842-200203000-00004. PMID 11914437
- [Background] Heale R, Forbes D. Understanding triangulation in research. Evid Based Nurs. 2013 Oct;16(4):98. doi: 10.1136/eb-2013-101494. Epub 2013 Aug 13. No abstract available. PMID 23943076
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hawkes AL, Hughes KL, Hutchison SD, Chambers SK. Feasibility of brief psychological distress screening by a community-based telephone helpline for cancer patients and carers. BMC Cancer. 2010 Jan 12;10:14. doi: 10.1186/1471-2407-10-14. PMID 20067645
- [Background] Hassanein KA, Musgrove BT, Bradbury E. Psychological outcome of patients following treatment of oral cancer and its relation with functional status and coping mechanisms. J Craniomaxillofac Surg. 2005 Dec;33(6):404-9. doi: 10.1016/j.jcms.2005.05.005. Epub 2005 Oct 25. PMID 16253509
- [Background] Harrop E, Noble S, Edwards M, Sivell S, Moore B, Nelson A. Managing, making sense of and finding meaning in advanced illness: a qualitative exploration of the coping and wellbeing experiences of patients with lung cancer. Sociol Health Illn. 2017 Nov;39(8):1448-1464. doi: 10.1111/1467-9566.12601. Epub 2017 Oct 16. PMID 29044627
- [Background] Greer S, Moorey S, Baruch JD, Watson M, Robertson BM, Mason A, Rowden L, Law MG, Bliss JM. Adjuvant psychological therapy for patients with cancer: a prospective randomised trial. BMJ. 1992 Mar 14;304(6828):675-80. doi: 10.1136/bmj.304.6828.675. PMID 1472184
- [Background] Greer S, Moorey S, Baruch J. Evaluation of adjuvant psychological therapy for clinically referred cancer patients. Br J Cancer. 1991 Feb;63(2):257-60. doi: 10.1038/bjc.1991.60. PMID 1997103
- [Background] Graves KD, Arnold SM, Love CL, Kirsh KL, Moore PG, Passik SD. Distress screening in a multidisciplinary lung cancer clinic: prevalence and predictors of clinically significant distress. Lung Cancer. 2007 Feb;55(2):215-24. doi: 10.1016/j.lungcan.2006.10.001. Epub 2006 Nov 3. PMID 17084483
- [Background] Goldberg DP, Blackwell B. Psychiatric illness in general practice. A detailed study using a new method of case identification. Br Med J. 1970 May 23;1(5707):439-43. doi: 10.1136/bmj.2.5707.439. PMID 5420206
- [Background] Glover J, Dibble SL, Dodd MJ, Miaskowski C. Mood states of oncology outpatients: does pain make a difference? J Pain Symptom Manage. 1995 Feb;10(2):120-8. doi: 10.1016/0885-3924(94)00073-t. PMID 7730684
- [Background] Gloster AT, Klotsche J, Chaker S, Hummel KV, Hoyer J. Assessing psychological flexibility: what does it add above and beyond existing constructs? Psychol Assess. 2011 Dec;23(4):970-82. doi: 10.1037/a0024135. Epub 2011 Jul 18. PMID 21767025
- [Background] Gellrich NC, Handschel J, Holtmann H, Kruskemper G. Oral cancer malnutrition impacts weight and quality of life. Nutrients. 2015 Mar 27;7(4):2145-60. doi: 10.3390/nu7042145. PMID 25825828
- [Background] Rouleau CR, Garland SN, Carlson LE. The impact of mindfulness-based interventions on symptom burden, positive psychological outcomes, and biomarkers in cancer patients. Cancer Manag Res. 2015 Jun 1;7:121-31. doi: 10.2147/CMAR.S64165. eCollection 2015. PMID 26064068
- [Background] Galway K, Black A, Cantwell M, Cardwell CR, Mills M, Donnelly M. Psychosocial interventions to improve quality of life and emotional wellbeing for recently diagnosed cancer patients. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD007064. doi: 10.1002/14651858.CD007064.pub2. PMID 23152241
- [Background] Franke GH, Jaeger S, Glaesmer H, Barkmann C, Petrowski K, Braehler E. Psychometric analysis of the brief symptom inventory 18 (BSI-18) in a representative German sample. BMC Med Res Methodol. 2017 Jan 26;17(1):14. doi: 10.1186/s12874-016-0283-3. PMID 28125960
- [Background] Foley E, Baillie A, Huxter M, Price M, Sinclair E. Mindfulness-based cognitive therapy for individuals whose lives have been affected by cancer: a randomized controlled trial. J Consult Clin Psychol. 2010 Feb;78(1):72-79. doi: 10.1037/a0017566. PMID 20099952
- [Background] Fiszer C, Dolbeault S, Sultan S, Bredart A. Prevalence, intensity, and predictors of the supportive care needs of women diagnosed with breast cancer: a systematic review. Psychooncology. 2014 Apr;23(4):361-74. doi: 10.1002/pon.3432. Epub 2013 Oct 28. PMID 24677334
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Fawzy FI, Fawzy NW, Arndt LA, Pasnau RO. Critical review of psychosocial interventions in cancer care. Arch Gen Psychiatry. 1995 Feb;52(2):100-13. doi: 10.1001/archpsyc.1995.03950140018003. PMID 7848046
- [Background] Faury S, Koleck M, Foucaud J, M'Bailara K, Quintard B. Patient education interventions for colorectal cancer patients with stoma: A systematic review. Patient Educ Couns. 2017 Oct;100(10):1807-1819. doi: 10.1016/j.pec.2017.05.034. Epub 2017 Jun 3. PMID 28602564
- [Background] Fallowfield L, Ratcliffe D, Jenkins V, Saul J. Psychiatric morbidity and its recognition by doctors in patients with cancer. Br J Cancer. 2001 Apr 20;84(8):1011-5. doi: 10.1054/bjoc.2001.1724. PMID 11308246
- [Background] Engel GL. The clinical application of the biopsychosocial model. J Med Philos. 1981 May;6(2):101-23. doi: 10.1093/jmp/6.2.101. No abstract available. PMID 7264472
- [Background] Edgar L, Rosberger Z, Collet JP. Lessons learned: Outcomes and methodology of a coping skills intervention trial comparing individual and group formats for patients with cancer. Int J Psychiatry Med. 2001;31(3):289-304. doi: 10.2190/U0P3-5VPV-YXKF-GRG1. PMID 11841126
- [Background] Duan Y, Wang L, Sun Q, Liu X, Ding S, Cheng Q, Xie J, Cheng ASK. Prevalence and Determinants of Psychological Distress in Adolescent and Young Adult Patients with Cancer: A Multicenter Survey. Asia Pac J Oncol Nurs. 2021 Mar 9;8(3):314-321. doi: 10.4103/2347-5625.311005. eCollection 2021 May-Jun. PMID 33850965
- [Background] Donovan KA, Jacobsen PB. Progress in the implementation of NCCN guidelines for distress management by member institutions. J Natl Compr Canc Netw. 2013 Feb 1;11(2):223-6. doi: 10.6004/jnccn.2013.0029. PMID 23411388
- [Background] Donovan KA, Grassi L, McGinty HL, Jacobsen PB. Validation of the distress thermometer worldwide: state of the science. Psychooncology. 2014 Mar;23(3):241-50. doi: 10.1002/pon.3430. Epub 2013 Nov 11. PMID 25160838
- [Background] Dobkin PL. Mindfulness-based stress reduction: what processes are at work? Complement Ther Clin Pract. 2008 Feb;14(1):8-16. doi: 10.1016/j.ctcp.2007.09.004. Epub 2007 Nov 13. PMID 18243937
- [Background] Diener E, Lucas RE, Scollon CN. Beyond the hedonic treadmill: revising the adaptation theory of well-being. Am Psychol. 2006 May-Jun;61(4):305-14. doi: 10.1037/0003-066X.61.4.305. PMID 16719675
- [Background] de Graeff A, de Leeuw JR, Ros WJ, Hordijk GJ, Blijham GH, Winnubst JA. Long-term quality of life of patients with head and neck cancer. Laryngoscope. 2000 Jan;110(1):98-106. doi: 10.1097/00005537-200001000-00018. PMID 10646723
- [Background] Dastan NB, Buzlu S. Psychoeducation intervention to improve adjustment to cancer among Turkish stage I-II breast cancer patients: a randomized controlled trial. Asian Pac J Cancer Prev. 2012;13(10):5313-8. doi: 10.7314/apjcp.2012.13.10.5313. PMID 23244155
- [Background] Daher M. Cultural beliefs and values in cancer patients. Ann Oncol. 2012 Apr;23 Suppl 3:66-9. doi: 10.1093/annonc/mds091. PMID 22628419
- [Background] Dabrowski M, Boucher K, Ward JH, Lovell MM, Sandre A, Bloch J, Carlquist L, Porter M, Norman L, Buys SS. Clinical experience with the NCCN distress thermometer in breast cancer patients. J Natl Compr Canc Netw. 2007 Jan;5(1):104-11. doi: 10.6004/jnccn.2007.0011. PMID 17239330
- [Background] Cutillo A, O'Hea E, Person S, Lessard D, Harralson T, Boudreaux E. The Distress Thermometer: Cutoff Points and Clinical Use. Oncol Nurs Forum. 2017 May 1;44(3):329-336. doi: 10.1188/17.ONF.329-336. PMID 29493167
- [Background] Creamer M, Bell R, Failla S. Psychometric properties of the Impact of Event Scale - Revised. Behav Res Ther. 2003 Dec;41(12):1489-96. doi: 10.1016/j.brat.2003.07.010. PMID 14705607
- [Background] Cramer H, Lauche R, Klose P, Lange S, Langhorst J, Dobos GJ. Yoga for improving health-related quality of life, mental health and cancer-related symptoms in women diagnosed with breast cancer. Cochrane Database Syst Rev. 2017 Jan 3;1(1):CD010802. doi: 10.1002/14651858.CD010802.pub2. PMID 28045199
- [Background] Costanzo ES, Lutgendorf SK, Mattes ML, Trehan S, Robinson CB, Tewfik F, Roman SL. Adjusting to life after treatment: distress and quality of life following treatment for breast cancer. Br J Cancer. 2007 Dec 17;97(12):1625-31. doi: 10.1038/sj.bjc.6604091. Epub 2007 Nov 13. PMID 18000503
- [Background] Cook SA, Salmon P, Dunn G, Holcombe C, Cornford P, Fisher P. A Prospective Study of the Association of Metacognitive Beliefs and Processes with Persistent Emotional Distress After Diagnosis of Cancer. Cognit Ther Res. 2015;39(1):51-60. doi: 10.1007/s10608-014-9640-x. PMID 25657483
- [Background] Clark D. 'Total pain', disciplinary power and the body in the work of Cicely Saunders, 1958-1967. Soc Sci Med. 1999 Sep;49(6):727-36. doi: 10.1016/s0277-9536(99)00098-2. PMID 10459885
- [Background] Chopra I, Kamal KM. A systematic review of quality of life instruments in long-term breast cancer survivors. Health Qual Life Outcomes. 2012 Jan 31;10:14. doi: 10.1186/1477-7525-10-14. PMID 22289425
- [Background] Chiou YJ, Chiu NM, Wang LJ, Li SH, Lee CY, Wu MK, Chen CC, Wu YS, Lee Y. Prevalence and related factors of psychological distress among cancer inpatients using routine Distress Thermometer and Chinese Health Questionnaire screening. Neuropsychiatr Dis Treat. 2016 Oct 25;12:2765-2773. doi: 10.2147/NDT.S118667. eCollection 2016. PMID 27822049
- [Background] Chirico A, Lucidi F, Mallia L, D'Aiuto M, Merluzzi TV. Indicators of distress in newly diagnosed breast cancer patients. PeerJ. 2015 Jul 21;3:e1107. doi: 10.7717/peerj.1107. eCollection 2015. PMID 26244115
- [Background] Chen PY, Chang HC. The coping process of patients with cancer. Eur J Oncol Nurs. 2012 Feb;16(1):10-6. doi: 10.1016/j.ejon.2011.01.002. Epub 2011 Mar 3. PMID 21376664
- [Background] Chaturvedi SK. Psychiatric oncology: Cancer in mind. Indian J Psychiatry. 2012 Apr;54(2):111-8. doi: 10.4103/0019-5545.99529. PMID 22988317
- [Background] Chambers SK, Foley E, Clutton S, McDowall R, Occhipinti S, Berry M, Stockler MR, Lepore SJ, Frydenberg M, Gardiner RA, Davis ID, Smith DP. The role of mindfulness in distress and quality of life for men with advanced prostate cancer. Qual Life Res. 2016 Dec;25(12):3027-3035. doi: 10.1007/s11136-016-1341-3. Epub 2016 Jun 17. PMID 27315118
- [Background] Cella DF, Jacobsen PB, Orav EJ, Holland JC, Silberfarb PM, Rafla S. A brief POMS measure of distress for cancer patients. J Chronic Dis. 1987;40(10):939-42. doi: 10.1016/0021-9681(87)90143-3. PMID 3611291
- [Background] Cash TF. Body image: past, present, and future. Body Image. 2004 Jan;1(1):1-5. doi: 10.1016/S1740-1445(03)00011-1. PMID 18089136
- [Background] Carlson LE, Angen M, Cullum J, Goodey E, Koopmans J, Lamont L, MacRae JH, Martin M, Pelletier G, Robinson J, Simpson JS, Speca M, Tillotson L, Bultz BD. High levels of untreated distress and fatigue in cancer patients. Br J Cancer. 2004 Jun 14;90(12):2297-304. doi: 10.1038/sj.bjc.6601887. PMID 15162149
- [Background] Carlson LE. Mindfulness-based interventions for coping with cancer. Ann N Y Acad Sci. 2016 Jun;1373(1):5-12. doi: 10.1111/nyas.13029. Epub 2016 Mar 9. PMID 26963792
- [Background] Bradt J, Dileo C, Grocke D, Magill L. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD006911. doi: 10.1002/14651858.CD006911.pub2. PMID 21833957
- [Background] Bidstrup PE, Johansen C, Mitchell AJ. Screening for cancer-related distress: Summary of evidence from tools to programmes. Acta Oncol. 2011 Feb;50(2):194-204. doi: 10.3109/0284186X.2010.533192. PMID 21231781
- [Background] Akechi T, Okamura H, Yamawaki S, Uchitomi Y. Predictors of patients' mental adjustment to cancer: patient characteristics and social support. Br J Cancer. 1998 Jun;77(12):2381-5. doi: 10.1038/bjc.1998.396. PMID 9649163
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21231781/